CLINICAL TRIAL: NCT03114189
Title: Effects of Ascending Warm Footbaths on Sleep Disturbances in Women Before Climacteric
Brief Title: Kneipp Water Applications for Insomnia
Acronym: KWAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Petra Klose, Director, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-7003-BO
Record Dates: First submitted 2016-11-08; First posted 2017-04-14 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Sleep Disturbance
Keywords: Sleep disturbance; footbath; Kneipp; care of sleep; sleep
MeSH Terms: conditions — Parasomnias

ARMS (2):
- Footbath, care of sleep (Active Comparator): Warm water (37°C) filled up to the level of the ankle. Water has to be heated up to 42°C and increased to the calf 's half height within 15 minutes.
  Information about wrong and correct behaviour.
  Interventions: Procedure: footbath; Behavioral: care of sleep
- Care of sleep (Active Comparator): Information about wrong and correct behaviour.
  Interventions: Behavioral: care of sleep

INTERVENTIONS:
Procedure: footbath
  Arms: Footbath, care of sleep
Behavioral: care of sleep

SUMMARY:
The purpose of this study is to ascertain whether warm footbathes are effective on sleep disturbances in women before climacteric.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 18 years
* Regularly recurring sleeping disease (not less then 2 times a week for minimum 3 month)

Exclusion Criteria:

* secundary sleeping disease
* Mental diseases which require therapy
* Medication: benzodiazepine,Z-drugs, barbiturat, antihistaminika, melatonin
* Severe comorbidity
* Gravidity
* Shift work
* Voyages (>3 times during the study)
* regulary application of Kneipp
* Participation on other studies to therapy sleeping diseases or stress

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-11; Primary Completion 2018-07 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Change of sleep quality | T1: At the beginning of intervention, T2: After 4 weeks of intervention, T3: 12 weeks after randomization
  Use Pittsburgh sleep quality index

CONTACTS AND LOCATIONS:
Locations (1):
- • Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen, Essen, Germany